CLINICAL TRIAL: NCT06678516
Title: The Effect of One Month of Intermittent Fasting on the Blood Microbiome in Healthy Volunteers
Brief Title: Intermittent Fasting on the Blood Microbiome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Maikel Petrus Peppelenbosch, prof. dr., Erasmus Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: NL85947.078.23
Record Dates: First submitted 2024-11-04; First posted 2024-11-07 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Healthy
Keywords: Intermittent fasting; The blood microbiome; Healthy volunteers
MeSH Terms: conditions — Intermittent Fasting

STUDY DESIGN:
Intervention Model Description: This study is a randomized, cross-over trial with healthy participants aged 18-65 years. Following random order, participants must go through two study periods: one month of intermittent fasting and ad libitum diet (no restrictions), respectively, with one month of washout period following the first study period before participants cross over to the second study period.
  Since the intervention is performing/not performing fasting, the participants cannot be blinded. The participants are instructed and guided through the interventions and before randomization will sign the PIF.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intermittent fasting (Experimental): One month of intermittent fasting.
  Interventions: Dietary Supplement: Intermittent fasting
- Ad libitum diets (No Intervention): One month of ad libitum diets (no fasting and/or restriction).

INTERVENTIONS:
Dietary Supplement: Intermittent fasting — Participants are asked to abstain from any form of fasting or calorie restriction in one month of the study (which is also a pre-fasting washout for those volunteers that might be performing forms of fasting before the study) and then start with one month of intermittent fasting, with daily fasting duration from 7:30 to 18:30. Food is abstained from during fasting, only water and zero-calorie drinks like black coffee and unsweetened tea are allowed.
  Other Names: OMIF
  Arms: Intermittent fasting

SUMMARY:
The investigators previously demonstrated that the gut microbiome can be remodeled by one month of intermittent fasting (OMIF) in healthy volunteers and animal models, with a notable alteration observed in its overall composition which could be linked to improvement in liver function. The blood microbiome, which mirrors the human ecosystem and includes all microbes mainly including bacteria, archaea, and viruses, is a new-identified human microbiome assessment tool that is assumed to be more stable and representative than the gut microbiome, with substantial potential for the diagnosis and prediction of liver cirrhosis and cancer. However, the effect of OMIF, which mimics lifestyle change typically advised in liver disease, on this blood microbiome remains elusive at best. The aim of this study is to explore whether OMIF remodels the composition and function of the blood microbiome in healthy volunteers, through a Randomized controlled cross-over trial, with secondary outcomes on the association of blood microbiome with the gut microbiome.

DETAILED DESCRIPTION:
The major proportion of human blood DNA is mainly released from host cells or unborn babies, which is often used either as a unique material in testing for genomic variants associated with genetic disorders like trisomy or as a potential candidate in the diagnostic and prognostic approach to unveiling many inflammatory diseases, especially cancer. Nevertheless, a substantial proportion (~1%) of human blood cell-free DNA is non-human origin. This fraction has gained relatively little attention hitherto. With the development of next generation sequencing technology and bioinformatic tools, the origin of these ignored DNA fragments can be identified by alternatively assigning these non-human DNAs to genome of various microorganisms: such analysis reveals that this DNA is a collection of microbiome sequences and includes archaea and other bacteria, viruses, fungi, and even eukaryotes. Subsequently, the value of analyzing these microbial DNAs was illustrated by the discovery that they create unique microbiome signatures that deconvolute healthy controls, patients with cancers even between different cancer types. Further research showed that blood microbiome may even also direct pathogenic roles, mediating the development of acute decompensation of cirrhosis, for instance.

It is suggested that the blood microbiome may be an internal (blood) niche of overall external microbiome from either gastrointestinal tract, lung tract, oral cavity, or skin sites etc. These external microbiomes can be entirety or partially (e.g., DNA and LPS) transferred into the circulation by different transfer mechanisms, explaining the high sensitivity and specificity of using blood microbiome signature in mirroring disease in these tissues and tract sites. A novel example is the translocation of the gut microbiome via intestinal barrier into circulation by diffusion or transport during nutrition absorption, which is showed to be much faster especially under the injury of intestinal integrity (e.g., chronic stress and metabolic disease). Nevertheless, whether the gastrointestinal (oral and fecal) microbiome serves as a major source in general for blood microbiome remains unexplored so far.

Intermittent fasting is a popular dietary concept because of its perceived healthy benefits to weight loss. As a non-pharmacological dietary intervention strategy, intermittent fasting has been widely studied due to its significant healthy effect and applied for improving metabolic disease (liver function and lipid levels) and chronic stress, through a mechanism closely associated with the remodeling of the gut microbiome. Given the effect of intermittent fasting on the gut microbiome, intermittent fasting remains as a powerful strategy in exploring the effect of lifestyle change on the blood microbiome and especially its relationship with the gut microbiome as well as other health-associated parameters. This can provide insights into the origin of blood microbiome and its potential in serving as biomarker for disease prediction and therapeutic targets.

In this randomized controlled cross-over trial, the investigators aim to test the effect of one month of intermittent fasting (OMIF) on the blood microbiome in healthy volunteers. The specific aims are to 1) determine the effect of OMIF in shaping the blood microbiome, especially archaea; 2) evaluate whether the blood microbiome is associated with the gut microbiome. The investigators hypothesize that OMIF can influence the overall composition and function of blood microbiome. the investigators also hypothesize that the level of some taxa is stable over time, irrespective of lifestyle change, age, and gender.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* 18.5 =< BMI < 25 kg/m2
* All genders are included.
* Have not fasted (go for a day without any food) for any amount of days in the month before the start of the study
* Being willing to provide App-derived movement data over the course of the study
* Participants are willing to and capable of providing written informed consent.

Exclusion Criteria:

* Regular use medications such as antibiotics, steroids, beta blockers, and adrenergic-stimulating agents (self-report)
* Regular use prebiotic and/or probiotics (self-report)
* Intake of antibiotic at least in previous 1 months (self-report)
* Daily consumption of >10 cigarettes, or >6 cups of coffee (the latter because of the effects on circadian rhythm). (self-report)
* Chronic diseases including type 2 diabetes, hypertension, fatty liver disease, cancer, or autoimmune disease (self-report and clinical chemistry)
* Internal diseases, including those of the gastrointestinal tract, lung, heart, vasculature, liver, and kidney (self-report and clinical chemistry)
* Eating disorder or unconventional eating habits (self-report)
* Have a clinically significant abnormality as measured by a blood test
* Participation in another study (self-report)
* Habit of performing regular fasting (self-report)
* Women: pregnancy and breastfeeding (self-report)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-01-10 (Estimated); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
Change in blood Archaea | One month
  Change in blood Archaea after OMIF versus ad libitum diets will be measured with shotgun sequencing technology.

SECONDARY OUTCOMES:
Change in blood bacteria | One month
  Change in blood bacteria after OMIF versus ad libitum diets will be measured with shotgun sequencing technology.
Changes in blood viruses | One month
  Changes in blood viruses after OMIF versus ad libitum diets will be measured with shotgun sequencing technology.
The relationship between the blood and gut microbiome | One month
  The gut microbiome taxa after OMIF versus ad libitum diets will be evaluated using shotgun sequencing technology. The relationship between the blood and gut microbiome will be determined using statistical testing.

OTHER OUTCOMES:
Change in BMI | One month
  Weight in kilograms and height in meters will be combined to report BMI in kg/m^2.
Change in systolic and diastolic blood pressure | One month
  Changes in both systolic and diastolic blood pressure after OMIF versus ad libitum diets will be assessed with a blood pressure monitor.
Changes in circulating concentrations of liver enzymes alanine transaminase, aspartate aminotransferase, gamma-glutamyl transferase and alkaline phosphatase | One month
  Measured in blood samples [units/L]
Changes in circulating concentrations of glucose, hemoglobin, fatty acids and cholesterol | One month
  Measured in blood samples [mmol/L]
Change in circulating concentration of creatinine | One month
  Measured in blood samples [units/L]
Change in steps walked | One month
  The number of average steps walked after OMIF versus ad libitum diet will be recorded using phone Health App.
Change in calorie intake | One month
  Changes in monthly calorie intake (kcal) will be converted from each food type recorded to compare the difference after OMIF versus ad libitum diets.

CONTACTS AND LOCATIONS:
Overall Officials: Maikel P Peppelenbosch, MD, PhD, Principal Investigator — Erasmus Medical Center; Maikel P Peppelenbosch, MD, PhD, Study Chair — Erasmus Medical Center
Locations (2):
- Northwest Minzu University, Lanzhou, Gansu, China
- Erasmus Medical Center - Department of Gastroenterology and Hepatology, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Su J, Hansen BE, Ma Z, Peppelenbosch MP. Effects of one month of intermittent fasting on the blood microbiome in healthy volunteers (OMIF): A randomized controlled crossover study protocol. Contemp Clin Trials. 2025 Aug;155:107986. doi: 10.1016/j.cct.2025.107986. Epub 2025 Jun 15. PMID 40527395